CLINICAL TRIAL: NCT04012593
Title: Single Centered Diary-based Study to Identify Course and Characteristics of Hormone Withdrawal Headaches/Migraines in Users of Combined Hormonal Contraceptives
Brief Title: Diary-based Study on the Course of Hormone-withdrawal Migraines
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01791
Record Dates: First submitted 2017-09-27; First posted 2019-07-09 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2019-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- premenopausal women: diary
  Interventions: Behavioral: Diary

INTERVENTIONS:
Behavioral: Diary

SUMMARY:
Single centered diary-based study to identify course and characteristics of hormone withdrawal headaches/migraines in users of combined hormonal contraceptives Objectives of the Research Project: to identify the course and characteristics of hormone withdrawal headaches/migraines in users of combined hormonal contraceptives (CHC)

DETAILED DESCRIPTION:
Participant recruitment is performed through advertisement placed in University Zürich (USZ) online. Advertisement in offices of neurologists and headache specialists, homepage of the Swiss headache society.

Interested women contact the investigators via email and are called back by one of the study doctors or students within 1 day from Monday-Friday. This phone call is thought to inform the women about the study in more detail and for the investigators to check eligibility. During this call the participants are informed about the study procedure and can ask any question. Here most important points are use of a CHC in a 21/7 regimen, regular (at least once on two months) withdrawal migraine/headaches, intention to continue the use of the contraceptive for 3 more months.

If the participants decide to participate, inclusion and exclusion criteria are checked. If women are applicable they receive the consent form and the study information with an envelope for return. If more questions come up the investigators are available per email and phone for answers. If a patient doesn't return the consent form the investigator will delete the personal data, which collected before. Only the year of birth will be noted in the personal data.

After consent participants receive headaches diaries (with mail /post) and a prepaid envelope (for return). Participants are also offered the option to return their diaries electronically via email to the study doctor. Furthermore participants receive in a second phone contact instructions, how to fill in the headache diary and the day of study start (first day of the next pill package).

Headache diaries should be returned monthly (per email or post) and are conducted for 3 pill cycles.

If complete headache diaries are not returned participants will be contacted per email after 1 week to remind the participants. If this email is not being answered within another week a phone contact will take place to identify potential reasons for noncompliance or withdrawal of consent or drop out.

Observation period 3 pill cycles : 3 times 28 days

Outcomes of the Research Project:

* Daily number of headaches and migraine in each day of the observation cycle.and during the Hormone-free interval (HFI)
* First day of migraine in the pill-free interval
* Start of migraine in relation to withdrawal bleeding
* Start of and number of prolonged migraines >24 hours in the pill-free interval and the phase of hormone intake.
* Pain intensity in the pill-free interval in comparison to the pill-phase
* Number of rescue medications/ migraine day during HFI and during pill intake
* efficacy of the medications (did medication stop the attack and did the attack return after maximal 8 hours)
* Within patient variability of the first migraine day in the HFI.

Statistical Methodology:

* Primary and secondary endpoints will be calculated as frequencies and percentages.
* For comparison the number of prolonged attacks during pill use and the HFI prolonged attacks per day of the observation interval are calculated and thereafter chi-square test for comparisons is used .
* Software programme is used for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Age 18-50 years
* Use of combined hormonal contraceptives 21/7 regimen
* Suffering from headache/migraine in the HFI.
* Women are allowed to use their normal headache medications

Exclusion Criteria:

* Withdrawal of consent
* incomplete diaries
* pregnancy
* migraine/headache in only 1 cycle
* inability to follow procedures (e.g. due to psychological disorders or dementia), insufficient knowledge of project language).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Premenopausal women
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Migraine in the pill-free interval | up to 3 months
  Migraine at each day of the pill-free interval

SECONDARY OUTCOMES:
First migraine day | up to 3 months
  First day of migraine in the pill-free interval
migraine episodes | up to 3 months
  Start of migraines >24 hours in the pill-free interval

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Merki, Professor, Study Director — University Hospital, Zürich
Locations (1):
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No